CLINICAL TRIAL: NCT01372475
Title: A Multi-Centre, Double-Blind, Randomized, Placebo Controlled Study To Evaluate The Safety And Effectiveness Of A New Viscoelastic Hydrogel (Hymovis) In The Treatment Of Knee OA With An Open-Label Extension
Brief Title: Hymovis™ Versus Placebo in Knee Osteoarthritis
Acronym: Hymovis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fidia Farmaceutici s.p.a. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R29-09-02
Record Dates: First submitted 2011-06-10; First posted 2011-06-14 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-03

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Knee; Hyaluronan; Hyaluronic Acid; Viscoelastic; Hydrogel
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hymovis Viscoelastic Hydrogel (Active Comparator): Intra-articular Injection
  Interventions: Device: Hymovis Intra-articular Injection
- Placebo (Placebo Comparator): Phosphate Buffered Saline Intra-articular Injection
  Interventions: Procedure: Phosphate Buffered Saline Injection

INTERVENTIONS:
Device: Hymovis Intra-articular Injection — Hymovis Intra-articular injection
  Other Names: HYADD4™; Hyaluronic Acid; HA; Hyaluronate
  Arms: Hymovis Viscoelastic Hydrogel
Procedure: Phosphate Buffered Saline Injection — Placebo Intra-articular injection
  Other Names: PBS; Saline
  Arms: Placebo

SUMMARY:
Purpose: The purpose of this study is to demonstrate if the intra-articular injection of a new viscoelastic Hydrogel (Hymovis) is superior to Placebo (phosphate buffered saline [PBS] in subjects with symptomatic osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ambulant outpatients ≥ 40 years of age with an active lifestyle:
2. Has a medical history of OA symptoms confirmed at least 3 months prior to the screening visit with radiographic evidence of OA, Kellgren-Lawrence grade 2-3
3. Discontinuation of any analgesic/NSAID therapy prior to baseline with no intent to resume during study

Exclusion Criteria:

1. Clinically significant apparent large effusion of the target knee;
2. Clinically significant valgus/varus deformities, ligamentous laxity or meniscal instability as assessed by the Investigator;
3. Any musculoskeletal condition affecting the target knee that would impair assessment of the effectiveness in the target knee such as Paget's disease
4. Medical history of anaphylactic reactions
5. History of septic arthritis in any joint
6. Females who are pregnant or breast-feeding

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2011-03; Primary Completion 2012-11 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Pain sub-score | 26 weeks
  WOMAC A Pain sub-score

SECONDARY OUTCOMES:
Responder Analysis | 26 weeks
  Outcome Measures in Rheumatoid Arthritis Clinical Trials - Osteoarthritis Research Society International (OMERACT-OARSI) Criteria
WOMAC Function | 26 Weeks
  WOMAC C Function sub-score
Visual Analog Scale (VAS) WOMAC Pain | 26 Weeks
  Question A1 of WOMAC Pain sub-score
WOMAC Global Score | 26 Weeks
WOMAC Stiffness sub-score | 26 Weeks
  WOMAC C stiffness sub-score
Rescue Medication Usage Pill Count, Failure Outcome | 26 Weeks
Patient Global Analysis | 26 Weeks
Clinician Responder Analysis | 26 Weeks
SF Health Outcome | 26 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Secchieri, PhD, Study Director — Fidia Farmceutici S.p.A.
Locations (33):
- United States (32):
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - Core Orthopaedic, Encinitas, California
  - San Diego Clinical Trials, San Diego, California
  - Norwalk Medical Group, Norwalk, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Tampa Bay Medical Research, Clearwater, Florida
  - Homestead Clinical Research, Cutler Bay, Florida
  - SJS Clinical Research, DeFuniak Springs, Florida
  - Avail Clinical Research, DeLand, Florida
  - Riverside Clinical Research, Edgewater, Florida
  - The Andrews Institute, Gulf Breeze, Florida
  - Sun Coast Clinical Research, New Port Richey, Florida
  - Pensacola Research Consultants, Pensacola, Florida
  - Lakeview Medical Research, Summerfield, Florida
  - Drug Studies America, Marietta, Georgia
  - Better Health Clinical Research, Newnan, Georgia
  - Sonora Clinical Research, Boise, Idaho
  - Rush University, Chicago, Illinois
  - Benchmark Research, Metairie, Louisiana
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Shores Rheumatology, Saint Clair Shores, Michigan
  - Columbus Clinical Research, Columbus, Ohio
  - Radiant Research, Columbus, Ohio
  - Blair Orthopedics Associates & Sports Medicine, Altoona, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - University Orthopedic Center, State College, Pennsylvania
  - Radiant Research, Anderson, South Carolina
  - Radiant Research, Greer, South Carolina
  - Tekton Research, Austin, Texas
  - Martin Diagnostic Center, Tomball, Texas
  - Orthopaedic Specialty Clinic, Spokane, Washington
- Latin Clinical Trial Center, San Juan, Puerto Rico